CLINICAL TRIAL: NCT03737253
Title: Clinical Study on Pharmacogenetics of Gonadotropin Receptors in Relation to Pregnancy and Life Birth Rate as Well as Unwanted Side Effects Such as Ovarian Hyper Stimulation Syndrome During Assisted Reproduction.
Brief Title: Hormone Evaluation in Artificial Reproductive Technology
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2016_467
Record Dates: First submitted 2018-10-23; First posted 2018-11-09 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Female Infertility
Keywords: gonadotropin; receptor; assisted reproduction
MeSH Terms: conditions — Infertility, Female | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa; follitropin beta; Urofollitropin; Menotropins

STUDY DESIGN:
Intervention Model Description: Women undergoing in vitro fertilization are allocated to either menotropin (urin derivate) or recombinant follicle stimulating hormone.
  Inclusion criteria are:
  * younger than 40 years of age
  * more than 12 months of unprotected intercourse
  * normal ovulatory cycles 26-32 days
  * first or second IVF treatment
  * indication for IVF is male factor
  * tubal factor or unexplained infertility.
  Exclusion criteria are:
  * Anti müllerian hormone less than 5pmol or FSH more than 12 cycle day 2-3
  * Endometriosis
  * polycystic ovarian syndrome
  * pre ovarian failure
  * smoking
  * male age more than 56.
  The succeeding treatment is according to normal procedures at respective clinic.
  End points are: total hormonal dosage, number of retrieved oocytes, fertilization rate, rate of blastocyst transfer, pregnancy rate, live birth rate.
  Adverse effects e.g overstimulation is recorded.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients and care providers need to know the type of hormone provided in order to be able to instruct and treat the patient. However, all roles are masked regarding the genotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Follitropin alpha (Active Comparator): Follitropin alpha (GONAL-f, Merck-Serono, Darmstadt, Germany), injections, dosage varying 1500-2500 IU, duration 2-5 days.
  Interventions: Drug: Follitropin alpha; Drug: Menotropin
- Menotropin (Active Comparator): Menotropin (Menopur, Ferring GmbH, Kiel, Germany), injections, dosage varying 1500-2500 IU, duration 2-5 days.
  Interventions: Drug: Follitropin alpha; Drug: Menotropin

INTERVENTIONS:
Drug: Follitropin alpha — The objective is to measure the effect of the drug according to gonadotropin receptor genotype.
  Other Names: Gonal F; Puregon; Urofollitropin
Drug: Menotropin — The objective is to measure the effect of the drug according to gonadotropin receptor genotype.
  Other Names: Menopur

SUMMARY:
The aim is to be able to predict the hormonal response according to gonadotropin receptor genotype and hormone type used for treatment of women undergoing in vitro fertilization or egg donation.

Outcome will be measured as pregnancy success, live born babies and unwanted side effects.

DETAILED DESCRIPTION:
Women undergoing in vitro fertilization receive high doses of the gonadotropins follicle stimulating hormone (FSH) and human chorionic gonadotropin (hCG), which is acting as luteinizing hormone (LH) for stimulation of the ovaries in order to obtain a high number of eggs. There are however marked individual differences in the hormonal response, ranging from lack of increased egg maturation to hyper stimulation. The hypothesis is that genetic variants in the gonadotropin receptors (LH and FSH receptors), are influencing the outcome. This assumption is supported by a recent study on more than 600 women undergoing in vitro fertilization, demonstrating that whereas only 10% of women with asparagine in both genes (FSHR N680S and LHR N312S) became pregnant, 40% of those with serine did (Lindgren I et al. Hum Repr 2016; 3:672-83).

Most (90%) of the women were treated with rFSH (recombinant). However, of the 10% asparagine carriers who actually became pregnant, most if not all, were treated with menotropin - a urine derivated compound (Menopur, Ferring), which contains both LH and FSH. This finding was not stressed in the manuscript as it could have been due to chance because of the small number of women treated with menotropin.

The objective is therefore to perform a prospective randomized study regarding efficacy of treatment in the first and second in vitro fertilization trial with rFSH and menotropin, respectively, genotype taken into account.

In total 890 women, 445 in Poznan, Poland and 445 in Malmö, Sweden, with unexplained infertility or a male or tubal factor indication for treatment will be invited to participate in the study. At first appointment, information is provided and informed consent retrieved. Two blood samples are drawn and stored at -20°C; one for subsequent genotyping and one for anti mullerian hormone measurement. The succeeding treatment is according to normal procedures at respective clinic.

ELIGIBILITY:
Inclusion Criteria:

* Normal ovulatory cycles 26-32 days
* First and second IVF treatment
* Indication for IVF is male factor, tubal factor or unexplained infertility
* Medical indication for IVF; >12 months unprotected intercourse

Exclusion Criteria:

* Anti Müllerian Hormone <5pmol or cycle day 2-3 FSH >12
* Endometriosis
* polycystic ovarian syndrome
* pre ovarian failure
* smoking
* male age more than 56.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 810 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Pregnancy | up to 12 months after treatment
  Association between pregnancy rate and genotype is evaluated

SECONDARY OUTCOMES:
Number of oocytes | up to 6 months after treatment
  Number of eggs developed in response to drug according to genotype is measured
live birth | up to 12 months after treatment
  Live birth rate according to genotype is analyzed

OTHER OUTCOMES:
Ovarian hyper stimulation syndrome | Up to 6 months after treatment
  Association between overreaction to hormonal stimulation and genotype is analysed
Poor response | Up to 6 months after treatment
  No or poor development of eggs in response to drug is analysed, genotype taken into account

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lundberg Giwercman, PhD, Principal Investigator — Lund University, Lund, Sweden
Locations (2):
- Poznan University of Medical Sciences, Poznan, Poland
- Reproductive Medicine Center, Malmo, Sweden